CLINICAL TRIAL: NCT03900884
Title: A Phase 1b Study of Palbociclib, Letrozole and Venetoclax in ER and BCL-2 Positive Locally Advanced or Metastatic Breast Cancer
Brief Title: Palbociclib, Letrozole & Venetoclax in ER and BCL-2 Positive Breast Cancer
Acronym: PALVEN
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18/028
Record Dates: First submitted 2019-04-01; First posted 2019-04-03 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Breast Neoplasm Female
MeSH Terms: interventions — venetoclax; palbociclib; Letrozole

STUDY DESIGN:
Intervention Model Description: This is a Phase 1b, open-label, multicentre dose escalation study of venetoclax in combination with palbociclib and letrozole in patients with ER positive and BCL-2 positive metastatic breast cancer. The study will enrol up to 36 patients with metastatic breast cancer, with the objective of defining the MTD of venetoclax in combination with palbociclib and letrozole. There will be up to a total of 6 dose levels. Three 'step-down' levels will also be included to incorporate the options of reducing the dose of palbociclib if required. The MTD will be the RP2D of palbociclib, letrozole and venetoclax.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Letrozole + Palbociclib + Venetoclax (Experimental): The Letrozole dose is 2.5 mg (D1-28) for all dose levels.
  Starting dose Level 1: Palbociclib 100 mg (D1-21) and Venetoclax 100 mg (D1-21) daily.
  Interventions: Drug: Venetoclax; Drug: Palbociclib; Drug: Letrozole

INTERVENTIONS:
Drug: Venetoclax — At commencement of study: Venetoclax will commence at 100 mg daily (oral) for days 1-21 of each 28 day cycle. This is a dose finding study so doses will be adjusted between 100 and 800 mg/day depending on dose escalation results and recommendation of the safety committee.
Drug: Palbociclib — At commencement of study: Palbociclib will commence at 100 mg daily (oral) for days 1-21 of each 28 day cycle. This is a dose finding study so doses will be adjusted between 75 and 125 mg/day depending on dose escalation results and recommendation of the safety committee.
Drug: Letrozole — Letrozole will be dosed daily at a fixed dose of 2.5 mg/day throughout the study.

SUMMARY:
This study is investigating the combination of palbociclib, letrozole and venetoclax in ER and BCL-2 positive locally advanced or metastatic breast cancer.

It is hypothesised that venetoclax may augment the actions of palbociclib and letrozole in these patient groups. The primary objective of the study is to determine the maximum tolerated dose of the combination treatment, which can be used in subsequent studies. The study will also investigate disease response and survival.

Participants will receive palbociclib (daily, on days 1-21 of each 28 day cycle), letrozole (daily, on days 1-28 of each 28 day cycle) and venetoclax (daily, on days 1-21 of each 28 day cycle) until the last patient has completed 18 months treatment on the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has provided written informed consent for the main PALVEN study.
2. Female patients ≥ 18 years of age at screening.
3. Postmenopausal, defined as:

   1. Age ≥60 years, or
   2. Age <60 years and undergone bilateral oophorectomy or medically confirmed ovarian failure, or
   3. Age <60 years and have cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause and have serum levels of oestradiol and FSH within the reference range for postmenopausal females.
4. If pre or peri menopausal, patients must be willing to receive ovarian suppression/ablation, commencing ≥28 days prior to first dose of treatment.
5. Eastern Cooperative Oncology Group (ECOG) performance status score ≤ 1. (Appendix 1).
6. Patient must have histological or cytological confirmation of metastatic carcinoma of the breast (either from the primary or metastatic site) or locally advanced breast cancer not amenable to surgical or local therapy with curative intent, with the following tumour molecular characteristics (as determined from pre-screening testing):

   1. ER positive (defined as ≥10% positive stained carcinoma cells).
   2. BCL-2 positive (defined as ≥50% cells with at least moderate cytoplasmic staining; intensity 2-3 on a 0-3 scale).
   3. HER2 non-amplified (per ASCO/CAP guidelines).
7. Patients must be willing to provide tissue after two weeks of treatment from a newly obtained core or excisional biopsy of a tumour lesion where feasible. Patients for whom a repeat biopsy cannot be provided (e.g. inaccessible or patient safety concern) may be eligible only upon agreement from the Coordinating Principal Investigator.
8. Patients have received no more than a total of two prior lines of systemic therapy for metastatic breast cancer. This can include one line of chemotherapy.
9. Patients must have measurable disease (according to RECIST v1.1) or evaluable disease. Bone-only metastases are allowed.
10. Patents must have adequate organ and bone marrow function as defined below within 14 days prior to registration:

    * Haemoglobin ≥ 90 g/L.
    * Absolute neutrophil count ≥ 1.5 x 109/L.
    * Platelet count ≥ 100 x 109/L.
    * ALT and AST ≤ 2.5 x upper limit of normal (ULN), or ≤ 5 x ULN if liver metastases are present.
    * Total serum bilirubin ≤ 1.5 x ULN. Patient's with Gilbert's syndrome may have a total serum bilirubin > 1.5 x ULN.
    * Creatinine Clearance ≥ 50 mls/min (Cockcroft-Gault, please see Appendix 2).
11. Female patients of childbearing potential must have negative urine or serum pregnancy test within 14 days prior to registration.
12. Life expectancy > 6 months.
13. Patient is able to swallow whole tablets.
14. Female patients of childbearing potential must be willing to use at least one of the following methods of contraception for the course of the study through to 30 days after the last dose of study medication:

    * Total abstinence from sexual intercourse as the preferred lifestyle of the patient (periodic abstinence is not acceptable).
    * Intrauterine device (IUD) or Mirena.
    * Double-barrier method (contraceptive sponge, diaphragm or cervical cap with spermicidal jellies or cream and a condom).

Exclusion Criteria:

1. Patients who have previously been exposed to venetoclax (ABT-199) or a CDK4/6 inhibitor (in the adjuvant or metastatic setting).
2. Patients who are pregnant or lactating.
3. Patients with evidence of CNS metastases.
4. Receipt of any anti-cancer therapy received within 21 days of registration including chemotherapy, radiotherapy, endocrine therapy (aromatase inhibitors, Selective Estrogen Receptor Modulator such as tamoxifen, or a Selective Estrogen Receptor Degrader such as fulvestrant) or other investigational therapy. The following therapies ARE permitted:

   1. Bisphosphonate or denosumab therapy for patients with bone metastases.
   2. Ovarian suppression in pre- and peri-menopausal patients.
5. Prior radiotherapy to a target lesion site, unless there has been unequivocal progression at that site following radiotherapy.
6. Patients who are taking warfarin or other oral anticoagulant therapy. The use of alternative anticoagulation therapy such as systemic low-molecular weight heparin will be acceptable.
7. Patients who have had major surgery within 28 days of first dose of study drug or anticipation of the need for major surgery during the course of study treatment.
8. Patients that have received any of the following agents within 7 days prior to registration:

   1. Steroid therapy for anti-neoplastic intent.
   2. CYP3A inhibitors e.g. fluconazole, ketoconazole, clarithromycin.
   3. Potent CYP3A inducers e.g. rifampicin, carbamazepine, phenytoin, St. John's Wort.
   4. Drugs that are known to prolong the QT interval (see Appendix 5).
9. Consumption of one or more of the following within 3 days prior to the first dose of study drugs:

   1. Grapefruit or grapefruit products.
   2. Seville oranges including marmalade containing Seville oranges.
   3. Star fruit (carambola).
10. Need for current chronic corticosteroid therapy (≥10 mg of prednisone per day or an equivalent dose of other corticosteroids).
11. Patients with active uncontrolled infection.
12. Patients with a known history of human immunodeficiency virus (HIV) infection, chronic Hepatitis B or C.

    1. Patients who are positive for HCV antibody must be negative for HCV by polymerase chain reaction (PCR) to be eligible.
    2. Patients with a post or resolved hepatitis B virus (HBV) infection (defined as having a positive HBcAb and negative HbsAg) may be included if HBV DNA is undetectable. These patients must be willing to undergo monthly DNA testing.
13. Administration of live, attenuated vaccine within 28 days prior to registration or anticipation of need for such a vaccine during the study.
14. Patients with a history of other malignancies within the past 5 years except for treated skin basal cell carcinoma (BCC), squamous cell carcinoma (SCC), malignant melanoma ≤1.0mm without ulceration, localised thyroid cancer, or cervical carcinoma in situ. Other malignancies considered to be at low risk of recurrence may also be included according to the discretion of the Investigator.
15. Patients with visceral spread at risk of short-term life-threatening complications.
16. Patients with a history of medical or psychiatric conditions that may interfere with the patient's participation in the study.
17. Patients on contraception that is oestrogen or progestin based (Mirena accepted).
18. Patients who are on Hormone Replacement Therapy.
19. Patients with a QTc ≥ 480 msec (based on the mean value of the triplicate ECGs), family or personal history of long or short QT syndrome, Brugada syndrome or known history of QTc prolongation, or Torsade de Pointes
20. Patients with an uncontrolled electrolyte disorder that can compound the effects of a QTc-prolonging drug (e.g. hypocalcemia, hypokalemia, hypomagnesemia)
21. History of a malabsorption syndrome or other condition that would interfere with enteral absorption of study drugs.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Determination of the Maximum Tolerated Dose (MTD), dose-limiting toxicities (DLTs) and recommended phase 2 dose of drug combination of palbociclib, letrozole and venetoclax. | 36 months
  To determine the MTD and DLTs of the combination of palbociclib, letrozole and venetoclax in ER positive, BCL-2 positive, HER2 negative metastatic breast cancer or locally advanced breast cancer not amenable to surgical or local therapy with curative intent, and to identify the recommended Phase 2 dose.

SECONDARY OUTCOMES:
Safety profile of the combination of palbociclib, letrozole and venetoclax: CTCAE V 5 | maximum 36 months
  Toxicities measured using CTCAE V 5
Response Rate | 24 weeks
  To describe the best response (according to RECIST v1.1), defined as Complete Response (CR) or Partial Response (PR) or stable disease (SD) at 24 weeks.
Overall survival | 36 months
  Overall survival (OS) defined as the time from commencement of the study to date of death from any cause
Clinical benefit rate | 36 months
  To estimate clinical benefit rate (CBR), defined as CR, PR or SD.
Patient reported outcomes | 36 months
  Defined as treatment-related symptoms, patient functioning, and health-related quality of life associated with venetoclax in combination with palbociclib and letrozole. Assessed through patient reported outcomes using a validated quality of life questionnaire - EORTC QLQ C30. The questionnaire is deigned to evaluate change in quality of life over time. Outcomes are rated by the patient on a numerical scale over 28 questions of between 1-4 With 1 being no issue to 4 being a significant issue. There are an additional 2 questions regarding overall quality of life which are rated on a numerical scale 1-7 with 1 being the poorest and 7 being excellent.

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Lindeman, MBBS FRACP PhD, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (3):
- Australia (3):
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Austin Health, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rodriguez Y, Unno K, Truica MI, Chalmers ZR, Yoo YA, Vatapalli R, Sagar V, Yu J, Lysy B, Hussain M, Han H, Abdulkadir SA. A Genome-Wide CRISPR Activation Screen Identifies PRRX2 as a Regulator of Enzalutamide Resistance in Prostate Cancer. Cancer Res. 2022 Jun 6;82(11):2110-2123. doi: 10.1158/0008-5472.CAN-21-3565. PMID 35405009
- [Derived] Muttiah C, Whittle JR, Oakman C, Lindeman GJ. PALVEN: phase Ib trial of palbociclib, letrozole and venetoclax in estrogen receptor- and BCL2-positive advanced breast cancer. Future Oncol. 2022 May;18(15):1805-1816. doi: 10.2217/fon-2021-1450. Epub 2022 Feb 21. PMID 35187951